CLINICAL TRIAL: NCT04067388
Title: Real Time Tissue Characterisation Using Mass Spectrometry
Brief Title: iKnife REIMS Project
Acronym: iKnife
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 124247
Record Dates: First submitted 2019-06-19; First posted 2019-08-26 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Neoplasms; Neoplasm Malignant
Keywords: iKnife; Mass sprectronomy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh ex vivo tissue samples for mass spectral (MS) analysis and histological examination where applicable (may be retained for long term storage and may be used in subsequent research including genetic testing, subject to having ethical approval)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rapid Evaporative Ionisation Mass Spectrometry (REIMS) — Use of iKnife instrument during standard operative practice

SUMMARY:
There are currently no widely accepted methods which provide real time in vivo, in situ tissue diagnostics within the operating theatre environment.

This project proposes that the oncological nature of in vivo tissue may be accurately identified using mass spectrometric analysis of tissue specific ions released during thermal degradation of tissue as occurs during electrosurgery.

Subsequently, the protocol describes a technique for a prospective study to determine whether Rapid Evaporative Ionisation Mass Spectrometry (REIMS) can be used to accurately identify the nature of human tissue both ex vivo and in vivo.

DETAILED DESCRIPTION:
The project aims/objectives comprise the following:

1. Building of histologically validated spectral databases for normal, benign and malignant tissue using ex vivo tissue analysis by Rapid Evaporative Ionisation Mass Spectrometry (REIMS).
2. Optimisation of a technique to provide accurate, real-time information on the nature of tissue intra-operatively using Rapid Evaporative Ionisation Mass Spectrometry.
3. Optimisation of a technique to provide accurate, real-time information on the nature of tissue during endoscopic procedures using Rapid Evaporative Ionisation Mass Spectrometry.
4. In vivo testing of the accuracy of the technique using pre-built spectral databases both intraoperatively and during endoscopic procedures including, but not limited to, the use of sub-study trials.
5. Validation of spectral data obtained using a second mass spectral analysis technique, Desorption Electrospray Ionisation Mass Spectrometry (DESI).
6. Bacterial identification from tissue using mass spectrometry, standard microbiology culture and metagenomic sequencing by '454 pyrosequencing.

The following will be collected from each enrolled participant:

1. Fresh ex vivo tissue samples for mass spectral (MS) analysis and histological examination where applicable
2. In vivo MS data from surgical diathermy smoke collected intra-operatively.

Custom built Mass spectrometers will be installed at participating sites. Optimal electrosurgical settings, in terms of obtaining maximal amount of good quality spectral data whilst providing adequate surgical dissection, will be determined between operating surgeons and researchers.

All spectral data collected will be uploaded anonymised into a research database with the full histology provided. The spectra will be pre-processed according to the mass spectrometer used for collection.

In addition to diagnostic accuracy REIMS offers additional advantages to existing and emerging IMA techniques. Specifically, the REIMS iKnife allows use of a standard operating procedure without altering operative workflow in that the technique samples the surgical aerosol already being generated during excision. The rapid time frame of analysis to results (1-2 seconds) means that eventually surgeons' decision-making may be altered in real-time to achieve negative margins or improve patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients who are able to provide informed consent
* Patients undergoing screening, endoscopy or surgical resection of tissue

Exclusion Criteria:

* All patients under the age of 18 years
* All patients who are pregnant
* Patients who are unable to provide informed consent or who do not wish to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing resectional surgery or gastrointestinal endocoscopic procedures.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Analysis of spectral data | 10 years
  To determine whether Rapid Evaporative Ionisation Mass Spectrometry (REIMS) can be used to accurately discern between cancerous and normal tissue both in vivo and ex vivo
Margin Analysis | 10 years
  The primary end-point is accuracy (sensitivity and specify) of rapid ionisation mass spectroscopy to distinguish between patients with at least one close or positive margin and those without close or positive margin.

SECONDARY OUTCOMES:
Tumour margin analysis | 10 years
  The primary end-point is accuracy (sensitivity and specify) of rapid ionisation mass spectroscopy to distinguish between patients with at least one close or positive margin and those without close or positive margin.

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan Takats, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Imperial College London, London
  - St. Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: No